CLINICAL TRIAL: NCT02819024
Title: Study of the Effects of Dexamethasone on Non-Small Cell Lung Cancer Using [F-18] FLT for Imaging With Positron Emission Tomography (PET)
Brief Title: Dexamethasone Effects in Patients With Refractory Non-Small Cell Lung Cancer Using FLT Positron Emission Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anthony F. Shields, MD PhD, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-174; NCI-2016-00881 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-174 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2016-06-20; First posted 2016-06-30 (Estimated); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dexamethasone, 18F-FLT PET) (Experimental): Patients receive dexamethasone PO BID on days 1-5. Patients undergo 3 18F-FLT PET scans. One scan within 7 days prior to the start of dexamethasone, one scan on day 3 after the 5th dose of dexamethasone, and one scan 6-9 days after the last dose of dexamethasone.
  Interventions: Drug: Dexamethasone; Device: Device for PET; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Dexamethasone — Given PO BID
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Device: Device for PET — Undergo 18F-FLT PET scan
  Other Names: 18F-FLT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; Fluorothymidine F 18; FLUOROTHYMIDINE F-18
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo 18F-FLT PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot research trial studies the effects of dexamethasone in patients with non-small cell lung cancer that has not responded after previous treatment. Drugs such as dexamethasone can affect how tumors grow and respond to treatments. Imaging tests, such as fluoro-L-thymidine (FLT) positron emission tomography , use a small amount of radioactive substance to show changes in tumor cells. Studying the effects of dexamethasone on lung tumors using FLT positron emission tomography may help doctors plan better treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of dexamethasone (Dex) treatment in patients with relapsed non-small cell lung cancer (NSCLC) using 3'-fluorothymidine (FLT) positron emission tomography (PET) as measured by changes in tumor maximum standardized uptake value (SUVmax).

SECONDARY OBJECTIVES:

I. Assess the reversibility of Dex-mediated changes in tumor FLT retention following the withdrawal of Dex.

II. Measure tumor Glucocorticoid Receptor alpha expression (GRα) from recent patient biopsy samples.

III. Analyze blood samples obtained during imaging to determine serum Dex concentration and for senescence markers in circulating tumor cells.

OUTLINE:

Patients receive dexamethasone orally (PO) twice daily (BID) on days 1-5. Patients undergo 3 fluorothymidine F-18 (18F)-FLT PET scans. One scan within 7 days prior to the start of dexamethasone, one scan on day 3 after the 5th dose of dexamethasone, and one scan 6-9 days after the last dose of dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven advanced non-squamous NSCLC. Patients may have newly diagnosed recurrent progressive or refractory disease which may be localized or wide spread.
* No chemotherapy for at least 4 weeks and no radiation to the index lesion or clear progression in that lesion (greater than 20% increase in longest diameter).
* Life expectancy of greater than 4 weeks
* Absolute neutrophil count >= 1,000/mcL (measured within 2 weeks of registration)
* No history of human immunodeficiency virus (HIV) or active infections
* No history of diabetes
* No surgery in the last 2 weeks prior to study enrollment
* Has not received Dex or another corticosteroid in over 4 weeks prior to enrollment
* Ability to understand and the willingness to sign a written informed consent document
* Agreed to FLT-PET imaging and signed consent and eligible FLT-PET protocol 2006-127
* Registered with the clinical trials office of the Karmanos Cancer Center/Wayne State University

Exclusion Criteria:

* Patients must have measureable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques (computed tomography [CT], magnetic resonance [MR] or PET); lesions in the previously irradiated area can be considered as measureable lesions as long as there has been an increase of at least 10 mm when compared to measurements obtained after completion of radiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06; Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Shields, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Wayne State University/Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Dexamethasone, 18F-FLT PET)
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Dexamethasone, 18F-FLT PET)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 63 [47 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor SUVmax Assessed by 18F-FLT PET Imaging
Description: The primary endpoint is reported with mean and standard deviation
Time Frame: Baseline to day 9
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | Treatment (Dexamethasone, 18F-FLT PET)
Number analyzed (Participants) | 5
SUVmax | -0.39 (0.39)
Statistical Analysis 1: Comparison: Treatment (Dexamethasone, 18F-FLT PET); Test type: Other; p = 0.087, t-test, 2 sided

2. Secondary Outcome: Fold Change in Senescence Marker Gro-alpha
Description: Fold change in senescence marker Gro-alpha from scan 1 to scan 3
Time Frame: Baseline to day 9
Measure: Mean (Standard Deviation); unit: fold change is unitless
Arm/Group | Treatment (Dexamethasone, 18F-FLT PET)
Number analyzed (Participants) | 2
fold change is unitless | 2.46 (0.35)

3. Secondary Outcome: Fold Change in Senescence Marker Gro-beta
Description: Fold change in senescence marker Gro-alpha from scan 1 to scan 3
Time Frame: Baseline to day 9
Measure: Mean (Standard Deviation); unit: fold change is unitless
Arm/Group | Treatment (Dexamethasone, 18F-FLT PET)
Number analyzed (Participants) | 2
fold change is unitless | 8.34 (7.05)

4. Secondary Outcome: Fold Change in Senescence Marker MCP-1
Description: Fold change in senescence marker Gro-alpha from scan 1 to scan 3
Time Frame: Baseline to day 9
Measure: Mean (Standard Deviation); unit: fold change is unitless
Arm/Group | Treatment (Dexamethasone, 18F-FLT PET)
Number analyzed (Participants) | 2
fold change is unitless | 14.8 (17.37)

5. Secondary Outcome: Tumor Glucocorticoid Receptor Alpha Expression
Time Frame: Baseline
Population: Needle biopsies were collected for routine care. There was not enough tissue left after the routine care analyses to perform the exploratory analysis specified in this endpoint.
Arm/Group | Treatment (Dexamethasone, 18F-FLT PET)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the date of informed consent until the 3rd scan 6~8 days after scheduled Dex treatment, an average of 5 weeks
Arm/Group | Treatment (Dexamethasone, 18F-FLT PET)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT02819024/Prot_SAP_000.pdf